CLINICAL TRIAL: NCT01946009
Title: A Prospective, With One Site, Open-label Not Controled Trial, for the Observation of Treatment With CIDOFOVIR 1%, 3 Nights Per Week, During 4 Weeks, of Anal Intraepithelial Neoplasia, High Level, in HIV+ Patients
Acronym: CIDAN12
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion SEIMC-GESIDA (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GESIDA-7412
Record Dates: First submitted 2013-03-21; First posted 2013-09-19 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2015-05

CONDITIONS: HIV
MeSH Terms: interventions — Cidofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cidofovir 1% (Experimental): Cidofovir 1% cream's basis, 2gr, three times per week, during 4 weeks.
  Interventions: Drug: Cidofovir 1% cream's basis, 2gr, three times per week, during 4 weeks.

INTERVENTIONS:
Drug: Cidofovir 1% cream's basis, 2gr, three times per week, during 4 weeks.

SUMMARY:
Cidofovir could be an effective drug for the treatment of Anal Intraepithelial Neoplasia(AIN).

ELIGIBILITY:
* Inclusion Criteria:

  1. Patients who have given informed consent in writing of the study before making any specific selection procedure for the study.
  2. Adult patients (18 years) with documented HIV infection, with high-grade AIN demonstrated by biopsy, and have not received any prior treatment for Anal Intraepithelial Neoplasia in the last 12 weeks.
  3. For women of childbearing potential, negative pregnancy test in urine screening visit. All women of childbearing age should continue effective contraception throughout the study treatment.
* Exclusion Criteria:

  1. Patients who have received previous treatment of Anal Intraepithelial Neoplasia (AIN) in the last 12 weeks. 2. Dermatoses in patients with anogenital area 3. Patients with a history of pre-invasive neoplasia associated with Human Papilloma Virus 4. Patients with a history of previous neoplasm, of any origin and location, in the past 5 years.

  5. Patients with a history of hematologic abnormalities, kidney or liver 6. Pregnant or breastfeeding women or women of childbearing age who do not wish to use adequate contraception at the discretion of the investigator.

  7. Any disease or condition of the patient which, in the opinion of the investigator, is not adequate patient participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with complete regression of anal intraepithelial neoplasia | 8 Weeks
  Describe the percentage of patients achieving complete regression of anal intraepithelial neoplasia (AIN), as confirmed by means of high-resolution anoscopy and biopsy

SECONDARY OUTCOMES:
Describe the percentage of patients that reduce the degree of Anal dysplasia | 8 weeks
  Describe the percentage of patients that reduce the degree of Anal dysplasia
Describe the percentage of patients that reduces the extent Intraepithelial Anal Dysplasia quadrants, although not complete regression | 8 Weeks
  Describe the percentage of patients that reduces the extent Intraepithelial Anal Dysplasia quadrants, although not complete regression
Time to relapse | 8 Weeks
  Describe the percentage of patients with recurrence after complete regression of HSIL and median time to relapse
Percentage of patients with clear of Human papillomavirus | 8 Weeks
  Describe the percentage of patients in whom Human Papillomavirus clears after treatment with cidofovir
Percentage of adverse events | 8 weeks
  Describe the number of patients with adverse events as a measure of safety and tolerability
Treatment effect | 8 Weeks
  Prospective Clinical Trial exploratory nature of the effect of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Elena Sendagorta, MD, Principal Investigator — Hospital La Paz
Locations (1):
- Hospital Universitario La Paz, Madrid, Spain

REFERENCES:
- [Derived] Sendagorta E, Bernardino JI, Alvarez-Gallego M, Feito M, Feltes R, Beato MJ, Perez-Molina JA, Yllescas M, Diaz-Almiron M, Arribas JR, Gonzalez-Garcia J, Herranz P; CIDAN127412 GESIDA Study Group. Topical cidofovir to treat high-grade anal intraepithelial neoplasia in HIV-infected patients: a pilot clinical trial. AIDS. 2016 Jan 2;30(1):75-82. doi: 10.1097/QAD.0000000000000886. PMID 26731755